CLINICAL TRIAL: NCT03967041
Title: Sarcopaenia is a Useful Risk Stratification Tool for Surgeons to Prognosticate Splenic Abscess Patients- A Retrospective Case Control Study
Brief Title: Sarcopaenia is a Useful Risk Stratification Tool for Surgeons to Prognosticate Splenic Abscess Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 106-4283C
Record Dates: First submitted 2019-05-20; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Splenic Abscess; Sarcopenia
Keywords: splenic abscess; sarcopenia; surgical emergency
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenic patients
  Interventions: Diagnostic Test: radiological defined sarcopenia
- Non-sarcopenic patients
  Interventions: Diagnostic Test: radiological defined sarcopenia

INTERVENTIONS:
Diagnostic Test: radiological defined sarcopenia — Evaluation for sarcopaenia was performed via calculating psoas cross-sectional area at level of L3 and normalising for height

SUMMARY:
Sarcopaenia is associated with poor prognoses of in-hospital mortality in splenic abscess patients. Investigators recommend its use by surgeons in the ED to rapidly risk stratify and identify patients requiring urgent and aggressive intervention, to maximise patient outcomes and survival chances.

DETAILED DESCRIPTION:
Splenic abscess is a life-threatening surgical emergency which requires early diagnosis and intervention to maximise patient outcomes. This can be achieved through accurate risk stratification in the emergency department (ED). Sarcopaenia refers to an age-related loss of skeletal muscle mass and strength with major physiologic and clinical ramifications. This study evaluates sarcopaenia as a radiological risk stratification tool to predict in-hospital mortality of splenic abscess patients.

99 adult patients at four training and research hospitals who had undergone abdominal contrast CT scans in the ED with the final diagnosis of splenic abscess from January 2005 to December 2015 were recruited. Evaluation for sarcopaenia was performed via calculating psoas cross-sectional area at level of L3 and normalising for height. Univariate analyses were used to evaluate the differences between survivors and non-survivors, with subsequent logistic regression analysis to assess odds ratio of sarcopaenia with respect to in-hospital mortality. A receiver operating characteristic (ROC) curve was plotted to determine predictability of sarcopaenia, with its corresponding sensitivity, specificity, and accuracy rate calculated.

ELIGIBILITY:
Inclusion Criteria:

All adult patients older than 20 years of age admitted to the aforementioned hospitals who had undergone an abdominal contrast CT scan in the ED with the final diagnosis of splenic abscess from January 2005 to December 2015

Exclusion Criteria:

Patients who could not be assessed for sarcopaenia in line with our study methodology and/or had other coexisting infections were excluded. Patients with abscesses involving the psoas muscles were also excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients visited emergency department with the diagnosis of splenic abscess
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 12 weeks
  In-hospital mortality during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided